CLINICAL TRIAL: NCT01047475
Title: A Phase II Trial of MB-6 Plus FOLFOX4 for Metastatic Colorectal Cancer
Brief Title: A Phase II Trial of MB-6 Plus FOLFOX4 for Metastatic Colorectal Cancer (FDA IND 103675)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB104CLCT01
Record Dates: First submitted 2009-12-22; First posted 2010-01-13 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
Keywords: MB-6; FOLFOX4; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MB-6+FOLFOX4 (Active Comparator): MB-6 6 capsules tid be taken with meals plus FOLFOX4, will be given for 16 weeks
  Interventions: Drug: MB-6
- Placebo+FOLFOX4 (Placebo Comparator): Placebo, 6 capsules tid be taken with meals plus FOLFOX4, will be given for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB-6 — 6# TID with meal
  Arms: MB-6+FOLFOX4
Drug: Placebo — 6# TID with meal
  Arms: Placebo+FOLFOX4

SUMMARY:
This is a randomized, double-blind, parallel group, placebo-controlled study evaluate the preliminary efficacy and safety of MB-6 (320 mg/capsule, 6 capsules tid) versus placebo in addition to standard chemotherapy in the treatment of patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed colorectal cancer and/or clinical evidence of metastasis;
2. At least one measurable lesion either by computer tomography (CT) scan or magnetic resonance imaging (MRI);
3. Aged 20 years old or above;
4. Eastern Cooperative Oncology Group (ECOG) performance status < 2;
5. Adequate bone marrow reserve (hemoglobin > 9 g/dl, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L);
6. Adequate renal and hepatic functions: total bilirubin < 1.25 x upper normal limit, creatinine < 1.25 x upper normal limit, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x upper normal limit;
7. Patients willing to participate in the trial and giving written informed consent.

Exclusion Criteria:

1. Pregnant or lactating patients;
2. Patients (male or female) with reproductive potential not using adequate contraceptive measures;
3. Patients with evidence of central nervous system metastasis;
4. Subject with active infection which requires systemic treatment of antibiotic, antifungal, or antiviral agents
5. Current history of chronic diarrhea;
6. Other serious illness or medical conditions (e.g.: history of angina, myocardial infarction);
7. History of second primary malignancies except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix;
8. Concurrent treatment with any other anticancer therapy;
9. Patients with congestive heart failure (New York Heart Association Functional Classification III or IV), epilepsy, or other significant medical conditions as judged by the investigator;
10. Patients treated with another investigational drug within 4 weeks of entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Chen, B.S., Principal Investigator — China Medical University Hospital
Locations (1):
- Microbio Co., Ltd., Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MB-6+FOLFOX4 | Placebo+FOLFOX4
Started | 34 | 38
Completed | 29 | 31
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB-6+FOLFOX4 | Placebo+FOLFOX4 | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 62.2 (13.71) | 63.0 (13.42) | 62.6 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  Taiwan | 34 | 38 | 72

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint of This Study is the Best Overall Response (Complete Response + Partial Response)
Description: The primary efficacy analysis, the incidence of best overall response during the study period, was based on the Fisher's exact test for the binary response that was used to test for the differences in the treatment efficacy between MB-6 and Placebo.
Time Frame: 16 weeks
Measure: Median (95% Confidence Interval); unit: percentage of Best overall Response
Arm/Group | MB-6+FOLFOX4 | Placebo+FOLFOX4
Number analyzed (Participants) | 34 | 38
percentage of Best overall Response | 61.76 [43.56 to 77.83] | 68.42 [51.35 to 82.50]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | MB-6+FOLFOX4 | Placebo+FOLFOX4
Serious Adverse Events (participants affected / at risk) | 6/34 | 13/38
Other Adverse Events (participants affected / at risk) | 34/34 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MB-6+FOLFOX4 (N=34) | Placebo+FOLFOX4 (N=38)
Neutropenia (Investigations) | 1 | 4
Pyrexia (General disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Device occlusion (Surgical and medical procedures) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Eteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematochezia (General disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Blood potassium decreased (Blood and lymphatic system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 1
Decreased appetite (General disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MB-6+FOLFOX4 (N=34) | Placebo+FOLFOX4 (N=38)
Neutropenia (Investigations) | 18 | 23
Platelet count decreased (Blood and lymphatic system disorders) | 21 | 20
Anaemia (Blood and lymphatic system disorders) | 12 | 20
Diarrhoea (Gastrointestinal disorders) | 14 | 18
Decreased appetite (General disorders) | 14 | 15
Aspartate aminotransferase increased (Hepatobiliary disorders) | 14 | 14
Fatigue (General disorders) | 13 | 14
Mucosal inflammation (General disorders) | 13 | 12
Nausea (Gastrointestinal disorders) | 13 | 11
Vomiting (General disorders) | 5 | 11
Alanine aminotransferase increased (Hepatobiliary disorders) | 9 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 7
White blood cell count decreased (Investigations) | 4 | 8
Blood creatinine increased (Investigations) | 2 | 7
Pyrexia (General disorders) | 4 | 4
Neutrophil count decreased (Investigations) | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5
Haemoglobin decreased (Blood and lymphatic system disorders) | 2 | 4
Hiccups (General disorders) | 3 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Oedema peripheral (General disorders) | 2 | 2
Weight decreased (General disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other